CLINICAL TRIAL: NCT00042068
Title: A Multi-center, Double-Blind, Randomized, Parallel-Group Trial to Compare the Efficacy and Safety of Three Doses of Meloxicam (7.5, 15, and 22.5 mg) and Placebo in Patients With Rheumatoid Arthritis
Brief Title: A Multi-Center Trial to Compare Three Doses of Meloxicam and Placebo in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 107.258
Record Dates: First submitted 2002-07-22; First posted 2002-07-24 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

INTERVENTIONS:
Drug: Meloxicam

SUMMARY:
A 12-week trial consisting of 5 visits (6 if follow up is needed) to find out how effective and safe three different doses of meloxicam are compared with placebo in Rheumatoid Arthritis. Patient will take one dose of study medication daily.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 and less than or equal to 80
* Diagnosis of Rheumatoid Arthritis for at least six weeks
* Taking an NSAID
* If female: using adequate contraception
* Willingness to stop current NSAID until criteria reached to begin study drug
* Able to provide written informed consent

Exclusion Criteria:

* Intolerance or hypersensitivity to NSAIDs or ingredients of trial drug
* Pregnancy, lactating
* Use of investigational drug within 30 days prior to entering the trial
* History of peptic ulcer or of gastrointestinal hemorrhage except simple hemorrhoidal bleeding
* History of cerebrovascular or other bleeding disorder
* Severe hypertension
* Other disease that might interfere with safety of the patient or evaluation of trial drug (investigator's opinion)
* RA of functional class IV
* Synovectomy in any large joint within the past 6 months prior to entering the trial or planned during trial
* Concomitant therapy with anticoagulant, therapeutic doses of aspirin, phenothiazines, lithium, chronic GI-medication, analgesic drug (except acetaminophen up to 4 grams/day)
* DMARDs initiated within past three months or dose changed less than two months before entering the trial
* Therapy with corticosteroids exceeding 10 mg/day prednisone equivalent or change in dose within 1 month before trial
* Concomitant therapy with ACTH within past month before entering the trial.
* History of narcotic or alcohol abuse (past 12 months)
* Abnormal laboratory values
* Previous participation in the present trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-06; Study Completion 2003-07

PRIMARY OUTCOMES:
Response according to American College of Rheumatology 20% (ACR20) classification | at 12 weeks

SECONDARY OUTCOMES:
Number of painful or tender joints | up to 12 weeks
Number of swollen joints | up to 12 weeks
Patient's global (overall) assessment of disease activity | up to 12 weeks
Investigator's global (overall) assessment of disease activity | up to 12 weeks
Patient's assessment of pain | up to 12 weeks
Patient's assessment of physical function (mHAQ) | up to 12 weeks
C-Reactive Protein (CRP) | up to 12 weeks
Withdrawal due to lack of efficacy | up to 12 weeks
Duration of morning stiffness | up to of 12 weeks
Patient's final global (overall) assessment of efficacy | at end of 12 weeks
Investigator's final global (overall) assessment of efficacy | at end of 12 weeks
Patient status with regard to change in arthritic condition | at end of 12 weeks
Use of rescue medication | up to 12 weeks
Incidence and intensity of adverse events | until 4 weeks post treatment
Patient's final global assessment of tolerability | at end of 12 weeks
Investigator's final global assessment of tolerability | at end of 12 weeks
Withdrawals due to adverse events | at end of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Ltd./Bracknell
Locations (148):
- United States (72):
  - Suites 570 (research) & 600 (PI), Huntsville, Alabama
  - Suite 200, Montgomery, Alabama
  - Suite 140, Anchorage, Alaska
  - #106, Glendale, Arizona
  - Suite 601, Phoenix, Arizona
  - Suite 201, Phoenix, Arizona
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Pasadena, California
  - Suite 100, Rancho Cucamonga, California
  - Boehringer Ingelheim Investigational Site, Rancho Mirage, California
  - Suite 208, San Diego, California
  - Suite 202, San Diego, California
  - Suite 301, San Leandro, California
  - Suite A, Santa Maria, California
  - Westlake Medical Research, Westlake Village, California
  - Suite 200, Colorado Springs, Colorado
  - Suites 205 & 206, Danbury, Connecticut
  - Suite 300, Washington D.C., District of Columbia
  - Boehringer Ingelheim Investigational Site, Delray Beach, Florida
  - Boehringer Ingelheim Investigational Site, Gainsville, Florida
  - Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - Boehringer Ingelheim Investigational Site, Largo, Florida
  - Suite 202, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Boehringer Ingelheim Investigational Site, Orlando, Florida
  - Suite 2, Orlando, Florida
  - Suite 406, Safety Harbor, Florida
  - Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - Boehringer Ingelheim Investigational Site, South Miami, Florida
  - Suite 101, St. Petersburg, Florida
  - Radiant Research, Stuart, Florida
  - Suite 203, Tampa, Florida
  - Boehringer Ingelheim Investigational Site, Zephyrhills, Florida
  - Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - Suite 202, Idaho Falls, Idaho
  - Boehringer Ingelheim Investigational Site, Lake Forest, Illinois
  - Boehringer Ingelheim Investigational Site, Rockford, Illinois
  - Boehringer Ingelheim Investigational Site, Springfield, Illinois
  - Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - Attn: Kathy Stoddard, Director, Wichita, Kansas
  - Suite 306, Wheaton, Maryland
  - Truesdale Clinic, Fall River, Massachusetts
  - Suite 202, Kalamazoo, Michigan
  - Suite 101, St Louis, Missouri
  - Suite 240, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, Lincoln, Nebraska
  - Boehringer Ingelheim Investigational Site, Reno, Nevada
  - PC, Jackson Commons D-2, Medford, New Jersey
  - Suite 8, Mercerville, New Jersey
  - Boehringer Ingelheim Investigational Site, New York, New York
  - Suite 100, Charlotte, North Carolina
  - Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - Boehringer Ingelheim Investigational Site, Camp Hill, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - Suite D, Mechanicsburg, Pennsylvania
  - Suite 331-333, Johnston, Rhode Island
  - Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - Suite H, North Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Orangeburg, South Carolina
  - Boehringer Ingelheim Investigational Site, Austin, Texas
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
  - Radiant Research, Dallas, Texas
  - Suite 200, Dallas, Texas
  - Suite 500, Lubbock, Texas
  - Suites 207, San Antonio, Texas
  - Suite 2A, Falls Church, Virginia
  - Boehringer Ingelheim Investigational Site, Everett, Washington
  - Suite D-3, Seattle, Washington
  - Boehringer Ingelheim Investigational Site, Yakima, Washington
- Argentina (2):
  - Boehringer Ingelheim Investigational Site, Buenos Aires
  - Boehringer Ingelheim Investigational Site, Rosario
- Australia (3):
  - Boehringer Ingelheim Investigational Site, Cotton Tree, Queensland
  - Emeritus Research, Malvern, Victoria
  - Department of Rheumatology, Perth, Western Australia
- Belgium (2):
  - Clinique du Parc Léopold, Brussels
  - Medisch Centrum van Huisartsen, Leuven
- Brazil (4):
  - Av Anhanguera 6479, Goiânia GO
  - Rua Ramiro Barcelos 2350, Porto Alegre RS
  - Boehringer Ingelheim Investigational Site, São Paulo - SP
  - Clínica de Doenças Parasitárias e Infecciosas-Hospital Dia, São Paulo - SP
- Canada (16):
  - 230-6091, Richmond, British Columbia
  - Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - Boehringer Ingelheim Investigational Site, Fort Erie, Ontario
  - Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - Dr. Denis O'Donnell, Kingston, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - Boehringer Ingelheim Investigational Site, Peterborough, Ontario
  - Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 104-532, St. Catharines, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Pointe-Claire, Quebec
- France (3):
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Nice
  - Boehringer Ingelheim Investigational Site, Tours
- Germany (13):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Augusta-Klinik, Bad Kreuznach
  - Boehringer Ingelheim Investigational Site, Bad Segeberg
  - Rheumatologie und Physikalische Therapie, Berlin
  - Boehringer Ingelheim Investigational Site, Ellefeld
  - Elisabeth-Krankenhaus, Essen
  - Boehringer Ingelheim Investigational Site, Klotten
  - ClinPharm International GmbH & Co. KG, Leipzig
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Steinhöring
  - Boehringer Ingelheim Investigational Site, Tübingen
  - Klinik für Rheumatologie,, Wiesbaden
- Hungary (9):
  - National Institute for Rheumatology and Physiotherapy, Budapest
  - DOTE, Debrecen
  - Aladár Petz County Hospital, Győr
  - St. Andrew State Hospital, Hévíz
  - St. Ferenc Hospital, Miskolc
  - Pál Almási Balogh Hospital, Ózd
  - Hungarian Brothers of St. John of Good, Pécs
  - Szegedi University, Szeged
  - Ferenc Csolnoky County Hospital, Veszprém
- Italy (4):
  - Università degli Studi, Genova
  - Ospedale Augusto Murri, Iesi
  - Università degli Studi di Napoli "Federico II", Napoli
  - Ospedale A. Galateo, SAN Cesario (Lecce)
- Russia (2):
  - Institute of Rheumatology of RAMN, Moscow
  - City Clinical Hospital No. 1, Moscow
- South Korea (5):
  - 896 Pyung Chon-Dong, Dongan-Gu, Gyeonggi-do
  - San-5, Woncheon-Dong, Paldal-Gu, Gyeonggi-do
  - 85 Jeo-Dong 2Ga, Seoul
  - Seoul National University Hospital, Seoul
  - Boehringer Ingelheim Investigational Site, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Rheumatology-Allergy-Immunology, Kaohsiung City
  - Chang Gung Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Ukraine (9):
  - Dnyepropyetrovsk Medical Academy, Dnyepropetrovsk
  - Central City Hospital, Donetsk
  - State Medical University, Donetsk
  - Municipal Institute of Health Care, Kharkiv
  - City Multitype Clinical Hospital No. 25, Kharkiv
  - Central Clinical Hospital, Kiev
  - Institute of Cardiology, Kiev
  - Regional Hospital No. 1, Kiev
  - Institute of Gerontology, Kyiv